CLINICAL TRIAL: NCT05355701
Title: A PHASE 1, OPEN-LABEL, DOSE ESCALATION AND DOSE EXPANSION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND ANTI TUMOR ACTIVITY OF PF-07799933 (ARRY-440) AS A SINGLE AGENT AND IN COMBINATION THERAPY IN PARTICIPANTS 16 YEARS AND OLDER WITH ADVANCED SOLID TUMORS WITH BRAF ALTERATIONS
Brief Title: A Study to Learn About the Study Medicine Called PF-07799933 in People With Advanced Solid Tumors With BRAF Alterations.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4761001; BRAF Class 2 (Other: Alias Study Number)
Record Dates: First submitted 2022-04-26; First posted 2022-05-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Melanoma; Non-Small-Cell Lung Cancer; Thyroid Cancer; Glioma; Advanced Colorectal Cancer (Part 1)
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Thyroid Neoplasms; Glioma | interventions — binimetinib; Cetuximab; Midazolam; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (9):
- Monotherapy dose escalation (Part 1) (Experimental): Participants will receive PF-07799933
  Interventions: Drug: PF-07799933
- Combination dose escalation (Part 2) (Experimental): Participants will receive PF-07799933 in combination with binimetinib or cetuximab
  Interventions: Drug: PF-07799933; Drug: binimetinib; Biological: cetuximab
- Dose expansion (Part 3) - Tumor and mutation specific Cohort 1 (Experimental): Participants will receive PF-07799933
  Interventions: Drug: PF-07799933
- Dose expansion (Part 3) - Tumor and mutation specific Cohort 2 (Experimental): Participants will receive PF-07799933
  Interventions: Drug: PF-07799933; Drug: binimetinib
- Dose expansion (Part 3) - Tumor and mutation specific Cohort 3 (Experimental): Participants will receive PF-07799933
  Interventions: Drug: PF-07799933; Drug: midazolam
- Dose expansion (Part 3) - Tumor and mutation specific Cohort 4 (Experimental): Participants will receive PF-07799933 in combination with cetuximab
  Interventions: Drug: PF-07799933; Biological: cetuximab
- Dose expansion (Part 3) - Tumor and mutation specific Cohort 5 (Experimental): Participants will receive PF-07799933 in combination with cetuximab and mFOLFOX6 regimen
  Interventions: Drug: PF-07799933; Biological: cetuximab; Drug: fluorouracil; Drug: leucovorin; Drug: oxaliplatin
- Dose expansion (Part 3) - Tumor and mutation specific Cohort 6 (Experimental): Participants will receive PF-07799933
  Interventions: Drug: PF-07799933
- Dose expansion (Part 3) - Tumor and mutation specific Cohort 7 (Experimental): Participants will receive PF-07799933
  Interventions: Drug: PF-07799933

INTERVENTIONS:
Drug: PF-07799933 — Tablet
  Other Names: ARRY-440
Drug: binimetinib — Tablet
  Other Names: Mektovi, PF-06811462, MEK162
  Arms: Combination dose escalation (Part 2); Dose expansion (Part 3) - Tumor and mutation specific Cohort 2
Biological: cetuximab — Injection for intravenous use
  Other Names: Erbitux
  Arms: Combination dose escalation (Part 2); Dose expansion (Part 3) - Tumor and mutation specific Cohort 4; Dose expansion (Part 3) - Tumor and mutation specific Cohort 5
Drug: midazolam — syrup
  Arms: Dose expansion (Part 3) - Tumor and mutation specific Cohort 3
Drug: fluorouracil — Injection for intravenous use
  Arms: Dose expansion (Part 3) - Tumor and mutation specific Cohort 5
Drug: leucovorin — Injection for intravenous use
  Arms: Dose expansion (Part 3) - Tumor and mutation specific Cohort 5
Drug: oxaliplatin — Injection for intravenous use
  Arms: Dose expansion (Part 3) - Tumor and mutation specific Cohort 5

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called PF-07799933) administered as a single agent and in combination with other study medicines in people with solid tumors.

This study is seeking participants who have an advanced solid tumor with a certain type of abnormal gene called "BRAF" and available treatments are no longer effective in controlling their cancer.

All participants in this study will receive PF-07799933. PF-07799933 comes as a tablet to take by mouth, 2 times a day. Depending on the part of the study, participants may also receive another study medicine:

* People with melanoma or other solid tumors may also receive binimetinib. Binimetinib comes as a tablet to take by mouth, 2 times a day.
* People with colorectal cancer may also receive cetuximab or cetuximab and mFOLFOX6 (Chemotherapy regimen). Cetuximab will be given weekly (or every two weeks) in the clinic as a shot given in the vein or port (intravenous, IV).

Participants may receive the study medicines for about 2 years. The study team will monitor how each participant is doing with the study treatment during regular visits at the study clinic.

ELIGIBILITY:
This study is seeking participants who meet the following key eligibility criteria:

Inclusion Criteria:

* Diagnosis of advanced/metastatic solid tumor including primary brain tumor.
* Qualifying BRAF alteration (V600 or non-V600 Class II/Class III BRAF alteration), in tumor tissue and/or blood (ie circulating tumor deoxyribonucleic acid [DNA], or ctDNA).
* Disease progressed during/following last prior treatment and no satisfactory alternative treatment options (Part 1, Part 2 (doublet), and Part 3 (cohorts 2, 3, 6, 7)).
* Tumor specific cohorts (melanoma, colorectal cancer) must have received specific prior approved therapies
* Part 3 (Cohort 1) (BRAF V600 mutant melanoma): Prior BRAF V600 inhibitor therapy required, prior MEK inhibitor therapy required, and immune checkpoint inhibitor therapy required.
* Part 3 (Cohort 4) (BRAF V600E CRC): Minimum of 2 cycles of prior 5-FU based chemotherapy required. No prior BRAF inhibitor/EGFR inhibitor allowed. Participants with MSI-H/dMMR mCRC should receive prior immune checkpoint inhibitor therapy.
* Part 3 (Cohort 5) (BRAF V600E CRC): No more than 2 cycles of prior 5-FU based chemotherapy allowed. No prior BRAF inhibitor/EGFR inhibitors allowed. Participants with MSI-H/dMMR mCRC should receive prior immune checkpoint inhibitor therapy.

Exclusion Criteria:

* Brain metastasis larger than 4 cm
* Systemic anti-cancer therapy or small molecule therapeutics ongoing at the start of study treatment.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO; history of retinal degenerative disease.
* Concurrent neuromuscular disorder associated with elevated creatine kinase (CK).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 267 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2028-11-02 (Estimated); Study Completion 2030-05-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLTs) (Part 1 and Part 2) | Cycle 1 (21 days)
  DLTs will be evaluated during the first cycle (21 days) as both a single agent or in combination with binimetinib or cetuximab
Number of participants with treatment-emergent adverse events (AEs) (Part 1 and Part 2) | Baseline to 28 days after last dose of study medication
  AEs as characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy
Number of participants with clinically significant change from baseline in laboratory abnormalities (Part 1 and Part 2) | Baseline to 28 days after last dose of study treatment
  Laboratory abnormalities as characterized by type, frequency, severity, and timing
Number of participants with clinically significant change from baseline in vital sign abnormalities (Part 1 and Part 2) | Baseline to 28 days after last dose of study treatment
  Vital sign abnormalities as characterized by type, frequency, severity, and timing
Dose interruptions due to AEs (Part 1 and Part 2) | Baseline to 2 years
  Incidence of dose interruptions due to AEs
Dose dose modifications due to AEs (Part 1 and Part 2) | Baseline to 2 years
  Incidence of dose modifications due to AEs
Discontinuations due to AEs (Part 1 and Part 2) | Baseline to 2 years
  Incidence of discontinuations due to AEs
Overall response rate (ORR) (Part 3) | Baseline to 2 years
  Response will be evaluated via radiographical tumor assessments by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Number of participants with clinically significant physical exam abnormalities (Part 1 and Part 2) | Baseline to 28 days after last dose of study treatment
  Physical exam abnormalities as as graded by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0

SECONDARY OUTCOMES:
Part 1 and Part 2: ORR | Baseline to 2 years
  ORR as assessed using the RECIST version 1.1.
Part 1/2/3: Intracranial response | Baseline to 2 years
  Intracranial response by RECIST version 1.1 (for brain metastases) & Response Assessment in Neuro-Oncology (RANO) - for primary brain tumors).
Part 1 and Part 2: Duration of response | Baseline to 2 years
  Duration of response
Part 3: Number of participants with treatment-emergent adverse events (AEs) | Baseline to 2 years
  AEs as characterized by type, frequency, severity, timing, seriousness, and relationship to study therapy
Part 3: Number of participants with clinically significant change from baseline in laboratory abnormalities | Baseline to 2 years
  Laboratory abnormalities as characterized by type, frequency, severity, and timing
Part 3: Number of participants with clinically significant change from baseline in vital sign abnormalities | Baseline to 2 years
  Vital sign abnormalities as characterized by type, frequency, severity, and timing
Part 3: Dose interruptions due to AEs | Baseline to 2 years
  Incidence of dose interruptions due to AEs
Part 3: Dose dose modifications due to AEs | Baseline to 2 years
  Incidence of dose modifications due to AEs
Part 3: Discontinuations due to AEs | Baseline to 2 years
  Incidence of discontinuations due to AEs
Part 3: Time to event endpoints in each combination | Baseline to 2 years
  Time to event endpoints in each combination
Part 3: Disease Control Rate (DCR) | Baseline to 2 years
  DCR
Part 1/2/3: PK parameters of PF-07799933, Single dose, maximum observed concentration (Cmax) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, Cmax
Part 1/2/3: PK parameters of PF-07799933, Single dose, time to maximum plasma concentration (Tmax) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, Tmax
Part 1/2/3: PK parameters of PF-07799933, Single dose, area under the plasma concentration-time curve from time 0 to the last time point of quantifiable concentration (AUClast) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, AUClast
Part 1/2/3: PK parameters of PF-07799933, Single dose, area under plasma concentration-time curve over 24 hours (AUC24) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, AUC24
Part 1/2/3: PK parameters of PF-07799933, Single dose, area under plasma concentration-time curve over 48 hours (AUC48) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, AUC48
Part 1/2/3: PK parameters of PF-07799933, Single dose, terminal elimination half life (t½) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, t½
Part 1/2/3: PK parameters of PF-07799933, Single dose, area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUCinf) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, AUCinf
Part 1/2/3: PK parameters of PF-07799933, Single dose, apparent oral clearance (CL/F) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, CL/F
Part 1/2/3: PK parameters of PF-07799933, Single dose, apparent volume of distribution (Vz/F) | Baseline to 2 years
  PK parameters of PF-07799933, Single dose, Vz/F
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, maximum observed concentration (Cmax) | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, Cmax
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, trough plasma or serum concentration (Ctrough) | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, Ctrough
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, time to maximum plasma concentration (Tmax) | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, Tmax
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, area under the plasma concentration-time curve over the dosing interval (AUCτ) | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, AUCτ
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, CL/F | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, CL/F
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, average plasma concentration (Cav) | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, Cav
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, peak-to-trough ratio (PTR) | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, PTR
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, accumulation ratio (Rac) | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, Rac (AUCτ /AUCsd,τ)
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, t1/2 | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, t1/2
Part 1/2/3: PK parameters of PF-07799933, Multiple dose, Vz/F | Baseline to 2 years
  PK parameters of PF-07799933, Multiple dose, Vz/F
Part 3: PK parameters of cytochrome P450 (CYP)3A4 probe substrate midazolam, Cmax | Baseline to 2 years
  PK parameters of CYP3A4 probe substrate midazolam, Cmax
Part 3: PK parameters of CYP3A4 probe substrate midazolam, Tmax | Baseline to 2 years
  PK parameters of CYP3A4 probe substrate midazolam, Tmax
Part 3: PK parameters of CYP3A4 probe substrate midazolam, AUClast | Baseline to 2 years
  PK parameters of CYP3A4 probe substrate midazolam, AUClast
Part 3: PK parameters of CYP3A4 probe substrate midazolam, t½ | Baseline to 2 years
  PK parameters of CYP3A4 probe substrate midazolam, t½
Part 3: PK parameters of CYP3A4 probe substrate midazolam, AUCinf | Baseline to 2 years
  PK parameters of CYP3A4 probe substrate midazolam, AUCinf
Part 3: PK parameters of CYP3A4 probe substrate midazolam, CL/F | Baseline to 2 years
  PK parameters of CYP3A4 probe substrate midazolam, CL/F
Part 3: PK parameters of CYP3A4 probe substrate midazolam, Vz/F | Baseline to 2 years
  PK parameters of CYP3A4 probe substrate midazolam, Vz/F
Part 3: TTR | Baseline to 2 years
  Time to response (TTR)
Part 3: DOR | Baseline to 2 years
  Duration of response (DOR)
Part 3: PFS | Baseline to 2 years
  Progression-free survival (PFS)
Part 3: OS | Baseline to 2 years
  Overall survival (OS)
Number of participants with clinically significant physical exam abnormalities (Part 3) | Baseline to 28 days after last dose of study medication
  Physical exam abnormalities as as graded by NCI CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (40):
- United States (31):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Highlands Oncology Group, Rogers, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Clinical and Translational Research Center (CTRC), Aurora, Colorado
  - UCHealth Sue Anschutz-Rodgers Eye Center, Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - University of Miami Sylvester Comprehensive Cancer Center-The Griffin Research Building, Miami, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - DFCI Chestnut Hill, Newton, Massachusetts
  - Brigitte Harris Cancer Pavilion, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - CT Scan and Echo Only: Henry Ford Medical Center-Plymouth, Plymouth, Michigan
  - MSK Monmouth, Middletown, New Jersey
  - MSK David H. Koch Center for Cancer Care, New York, New York
  - Memorial Sloan Kettering Cancer Center 53rd street, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic Taussig Cancer Center Investigational Pharmacy, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - TriStar Bone Marrow Transplant, Nashville, Tennessee
  - TriStar Centennial Medical Center - Cell Processing Lab, Nashville, Tennessee
  - TriStar Centennial Medical center, Nashville, Tennessee
  - START San Antonio, San Antonio, Texas
- Canada (5):
  - Cross Cancer Institute, Edmonton, Alberta
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- Israel (4):
  - Sheba Medical Center, Ramat Gan, Central District
  - Sourasky Medical Center, Tel Aviv, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Rambam Health Care Campus, Haifa, Ḥeifā

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4761001